CLINICAL TRIAL: NCT05437601
Title: Effect of Astaxanthin in Reducing Disease Activity in Moderate to Severe Knee Osteoarthritis: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effect of Astaxanthin in Moderate to Severe Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Masuma Tabassum, Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2022/5680
Record Dates: First submitted 2022-06-27; First posted 2022-06-29 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — astaxanthine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either 12 mg astaxanthin capsules or placebo capsules for 8 weeks
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will not know which arm patients have been assigned to or if they receive placebo or astaxanthin
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astaxanthin (Experimental): Patients will receive three capsules of astaxanthin (4mg) daily for 8 weeks.
  Interventions: Drug: Astaxanthin Oral Capsule
- Control (Placebo Comparator): Patients will receive three capsules of placebo daily for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Astaxanthin Oral Capsule — 12 mg oral astaxanthin daily for 8 weeks
  Other Names: 3,3'-dihydroxy-4,4'-diketo-β-β carotene,
  Arms: Astaxanthin
Other: Placebo — Oral placebo identical to astaxanthin
  Arms: Control

SUMMARY:
This study will be 8 weeks randomized, double-blind, placebo-controlled trail to assess the effect of astaxanthin in 80 moderate to severe knee osteoarthritis patients. Participants will be assessed at baseline and after 8 weeks of intervention. Subjects will be randomized to receive either astaxanthin 12 mg capsule daily or placebo capsule identical to astaxanthin daily for 8 weeks. Evaluation of pain, stiffness and improvement of physical function will be measured by WOMAC index before and after intervention. Inflammatory markers serum IL-6 and hsCRP will be measured before and after intervention. Astaxanthin related adverse events will be identified. Study outcome will establish safety and efficacy of astaxanthin in knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the leading cause of disability worldwide and knee is the commonest joint involved. In 2020 there were around 654.1 million individuals (40 years and older) with knee OA and this prevalence tend to increase rapidly due to the growing aging of the population as well as an increase in risk factors particularly obesity and sedentary lifestyle. Evidences show that OA is associated with chronic low grade inflammation. Nonsteroidal anti-inflammatory drugs (NSAIDs) are the mainstay of management for OA symptoms which however cause serious gastrointestinal, renal and cardiovascular adverse events. With the lack of safe and effective therapies for OA, many patients are eventually faced with costly total joint replacement as the only option to improve pain, function, and quality of life. Astaxanthin is a natural oxycarotenoid which exhibits strong anti-inflammatory and anti-oxidant effects and is a promising therapeutic potential in OA. Till date sufficient data is not available regarding effects of astaxanthin in OA in human. This study is an effort to explore whether astaxanthin as add on therapy with conventional treatment of OA produce improvement in disease activity and inflammatory indicators in moderate to severe knee OA patients. This study will be a randomized, double-blind, placebo-controlled trial and will be conducted in the Department of Pharmacology, BSMMU in collaboration with the Department of Physical Medicine and Rehabilitations, BSMMU. A total of eighty (80) OA patients attended in the outpatient Department of Physical Medicine and Rehabilitations, BSMMU will be selected for the study according to inclusion and exclusion criteria. Diagnosis of moderate and severe knee OA will be made radiologically by an expert physiatrist of Department of Physical Medicine and Rehabilitations, BSMMU using the Kellgren-Lawrence grading scale. Each participant will be assessed by translated and validated Bangla version of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) VA3.01 in a calm place in the BSMMU campus for pain, stiffness and physical function. Serum Interleukin-6 (IL-6) and high sensitive C-reactive protein (hsCRP) will be measured. Then participants will randomly be assigned into two groups: Intervention group and Control group. The intervention group patients will receive conventional treatment with astaxanthin 3 capsules of 4mg after breakfast daily for 8 weeks making a total dose of 12 mg astaxanthin/day. On the other hand, patients in control group will receive 3 placebo capsules of 4 mg after breakfast daily for 8 weeks along with conventional treatment given by the physiatrist. The regularity of medicine intake will be ensured over telephone, capsule count and from the patient's compliance sheet. After 8 weeks of therapy each participant will be assessed once again by Bangla version of WOMAC Index and serum IL-6 and hsCRP will be measured. Patients will be asked to inform if they encountered any astaxanthin related adverse events. Study outcomes will provide evidence to support astaxanthin's safety and efficacy as an added strategy for symptom management in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee pain
* Radiographic evidence of moderate to severe knee osteoarthritis
* Age 40 years or older
* Both male and female

Exclusion Criteria:

* Prior history of knee trauma or surgery
* Previously diagnosed of systemic inflammatory conditions such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease
* Known allergy to fish or astaxanthin
* Currently taking immunosuppressant
* Pregnant and nursing mother
* Patients unwilling to participate or unwilling to give written consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Effect of astaxanthin on Improvement of pain, stiffness and physical function | 8 weeks
  The investigators will address this by conducting a prospective, double-blinded, randomized, placebo-controlled trial in which 80 patients who have been diagnosed with moderate to severe osteoarthritis of the knee will randomly receive a 8-week oral daily course of either astaxanthin (12 mg) or placebo. Improvement of pain, stiffness and physical function will be measured by translated and validated Bangla version of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)

SECONDARY OUTCOMES:
Serum IL-6 | 8 weeks
  will be measured by commercially available ELISA kits before and after intervention
High sensitive C-reactive protein | 8 weeks
  will be measured before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Masuma Tabassum, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh